CLINICAL TRIAL: NCT02834286
Title: Low-dose Rituximab in Combination With Eltrombopag and High-dose Dexamethasone as Frontline Treatment for Immune Thrombocytopenia
Brief Title: Rituximab, Eltrombopag and Dexamethasone as Frontline Treatment for Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Hematology division chief, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE14-021
Record Dates: First submitted 2016-07-01; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; eltrombopag; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab, eltrombopag and dexamethasone (Experimental): Each patient will receive Rituximab 100 mg weekly days 1, 7, 14, 21 Eltrombopag 50 mg PO days 1-28 Dexamethasone 40 mg IV/PO days 1-4
  Interventions: Drug: Rituximab; Drug: Eltrombopag; Drug: Dexamethasone

INTERVENTIONS:
Drug: Rituximab — Rituximab 100 mg weekly days 1, 7, 14, 21
Drug: Eltrombopag — Eltrombopag 50 mg PO days 1-28
Drug: Dexamethasone — Dexamethasone 40 mg IV/PO days 1-4

SUMMARY:
The purpose of this study is to determine the response rate and response duration with the combination of low-dose rituximab, eltrombopag and high-dose dexamethasone.

DETAILED DESCRIPTION:
Immune thrombocytopenia is an autoimmune disorder characterized by formation of autoantibodies against platelet antigens leading platelet destruction.

Corticosteroids increase the platelet count in about 80 percent of patients. However, many patients have a relapse when the dose of corticosteroid is reduced. Debilitating side effects are common in patients who require long-term corticosteroid therapy to maintain the platelet count. Eltrombopag, it is a small molecule agonist of the c-mpl (TpoR) receptor, which is the physiological target of the hormone thrombopoietin, has been shown to be effectively raise the platelet count in adult patients (aged 18 years and over) who have had their spleen removed or where splenectomy is not an option and have received prior treatment with corticosteroids or immunoglobulins, and these medicines did not work (refractory ITP). There are a few case reports where eltrombopag was an option as first line treatment for IT.

The purpose of this study is to determine the response rate and response duration with the combination of rituximab (100 mg weekly four weeks), eltrombopag (50mg PO once a day, day 1-28) and high-dose dexamethasone (40mg PO days 1-4) in untreated adult patients with <30*109/L platelet count diagnosed with immune thrombocytopenia.

A complete response is defined as an increase in platelet counts to >150×109/L on two consecutive occasions. A clinical response is defined as an increase in the platelet count between >30×109/L on two consecutive measures and no bleeding. Duration of response is considered from the day of the initial administration to the first time of relapse (platelet count <30×109/L) or to time of analysis Patients will be evaluated each week during 4 weeks and then every month for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed immune thrombocytopenic (IT) Platelet count less than 30,000/mm3 on two ocasionts with bleeding.
* Subject ≥ 16 years
* Subject has signed and dated written informed consent.
* No sepsis or fever or active infection
* Not pregnant or nursing

Exclusion Criteria:

* Previous treatment (only corticosteroids at dose or prednisone equivalent of 300 mg)
* Performance status above or equal to 2.
* Pregnancy and lactation
* Previous splenectomy
* Connective tissue disease
* Autoimmune hemolytic anemia
* Relapse

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Response | 28 days
  Platelet counts to >30×109/L on two consecutive occasions

SECONDARY OUTCOMES:
Complete Response | 28 days
  Platelet counts to >100×109/L on two consecutive occasions

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Hematología, Hospital Universitario "Dr. José Eleuterio González", Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Gonzalez-Lopez TJ, Alvarez-Roman MT, Pascual C, Sanchez-Gonzalez B, Fernandez-Fuentes F, Jarque I, Perez-Rus G, Perez-Crespo S, Bernat S, Hernandez-Rivas JA, Andrade MM, Cortes M, Gomez-Nunez M, Olivera P, Martinez-Robles V, Fernandez-Rodriguez A, Fuertes-Palacio MA, Fernandez-Minano C, de Cabo E, Fisac R, Aguilar C, Barez A, Penarrubia MJ, Garcia-Frade LJ, Gonzalez-Porras JR. Eltrombopag safety and efficacy for primary chronic immune thrombocytopenia in clinical practice. Eur J Haematol. 2016 Sep;97(3):297-302. doi: 10.1111/ejh.12725. Epub 2016 Jan 27. PMID 26709028
- [Result] Kim YK, Lee SS, Jeong SH, Ahn JS, Yang DH, Lee JJ, Kim HJ. Efficacy and safety of eltrombopag in adult refractory immune thrombocytopenia. Blood Res. 2015 Mar;50(1):19-25. doi: 10.5045/br.2015.50.1.19. Epub 2015 Mar 24. PMID 25830126
- [Result] Gomez-Almaguer D, Herrera-Rojas MA, Jaime-Perez JC, Gomez-De Leon A, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Tarin-Arzaga L, Hernandez-Reyes J, Ruiz-Arguelles GJ. Eltrombopag and high-dose dexamethasone as frontline treatment of newly diagnosed immune thrombocytopenia in adults. Blood. 2014 Jun 19;123(25):3906-8. doi: 10.1182/blood-2014-01-549360. Epub 2014 May 6. PMID 24802773
- [Result] Gomez-Almaguer D, Tarin-Arzaga L, Moreno-Jaime B, Jaime-Perez JC, Ceballos-Lopez AA, Ruiz-Arguelles GJ, Ruiz-Delgado GJ, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Sanchez-Cardenas M. High response rate to low-dose rituximab plus high-dose dexamethasone as frontline therapy in adult patients with primary immune thrombocytopenia. Eur J Haematol. 2013 Jun;90(6):494-500. doi: 10.1111/ejh.12102. Epub 2013 Apr 2. PMID 23470153